CLINICAL TRIAL: NCT02462785
Title: Carbohydrate Counting and Type 1 Diabetes: A Randomized Controlled Trial of Internet-based Teaching for Adolescents Learning to Count
Brief Title: An Evaluation of Internet-based Carbohydrate Counting Education for Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Jill Hamilton, Senior Associate Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000042623
Record Dates: First submitted 2015-05-12; First posted 2015-06-04 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Adolescents; Carbohydrate Counting; Glycemic Control; Self-Management; T1DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-Class Instruction (Active Comparator): This group of adolescents will receive carbohydrate counting instruction through an in-person, in class session led by a registered dietician. This represents the usual standard of care at the Diabetes Clinic at The Hospital for Sick Children (SickKids).
  Interventions: Behavioral: In-person Carbohydrate Counting Class
- Internet-Based Teaching (Experimental): This group of adolescents will receive carbohydrate counting instruction through an online teaching tutorial.
  Interventions: Behavioral: Online Carbohydrate Counting Tutorial

INTERVENTIONS:
Behavioral: In-person Carbohydrate Counting Class — An in-person carbohydrate counting class led by a registered dietician. The in class session covers topics including the role of CHO in nutrition and diabetes, sources of CHO, different CHO and non-CHO foods, resources for CHO counting, label reading, and meal planning. This is the standard procedure for CHO counting education at SickKids.
  Arms: In-Class Instruction
Behavioral: Online Carbohydrate Counting Tutorial — A web-based CHO counting tutorial that covers the same concepts reviewed during the standard in-person instructional session held at SickKids. A teen delivers the educational messages in short segments using techniques designed to maintain the viewer's attention (e.g., visuals of food portions and short segment highlights to emphasize important points). The online module includes brief interactive question/answer components for reinforcement. The secure online tutorial will be accessible for one week through a link provided by REDCap. Users will be able to repeat sessions, log on and off during sessions, and choose specific modules for repetition/review. The investigators will be able to capture the number of times patients log on and detail frequency and specifics of usage.
  Arms: Internet-Based Teaching

SUMMARY:
Helping individuals with diabetes to control their blood sugars through self-management is an important goal, and counting carbohydrates (CHO) remains a key part of diabetes education and management. There is very little research examining CHO counting education with adolescents who have type 1 diabetes (T1DM). The purpose of this pilot study is to evaluate a newly developed internet-based teaching module of CHO counting for adolescents, ages 12-17 years, with T1DM and who do not regularly CHO count and require instruction. A secondary aim is to assess feasibility for a future, larger-scale clinical trail. An effective web-based CHO counting tutorial could be used to strengthen current diabetes education programs and may serve as a basis for developing other teaching modules. Advantages of web-based teaching include convenience, increased accessibility, and the ability to review and reinforce teaching concepts through repetition. It may also encourage adolescents to take the initiative for their own diabetes care, beginning with a self-directed, active learning experience.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-17 years with a diagnosis of T1DM for more than 1 year
* Followed at the SickKids Diabetes Clinic
* Have access to a computer with Internet connection
* Able to communicate in English

Exclusion Criteria:

* Patients with type 2 diabetes, medication-induced diabetes or other forms of non T1DM
* Patients with Celiac disease, due to differences in prescribed dietary regimen
* Patients who are unable to communicate in English
* No computer or internet access
* Patient with cognitive delay impeding their ability to learn CHO counting
* Patients who have attended a CHO counting class within the past 6 months
* Patients who do not eat the foods presented on the planned meal & snack trays

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Carbohydrate Counting Accuracy Measured Using a Standardized Meal & Snack Tray Test at Baseline and 3-months Post-Education | Baseline; 3-months post-education
  Test trays will comprise foods commonly consumed by adolescents (e.g., hamburger, grilled cheese sandwich). CHO counting accuracy using food trays will be checked against a computerized food analysis. Several tray combinations will be used with randomization to tray order within each group for both pre- and post- assessments.

SECONDARY OUTCOMES:
Change in Carbohydrate Counting Knowledge Tested Using the PedCarbQuiz (PCQ) at Baseline and 3-months Post-Education | Baseline; 3-months post-education
  A 52 item assessment of carbohydrate and insulin dose calculating knowledge in youth with T1DM

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton, MD, M.Sc., Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada